CLINICAL TRIAL: NCT04683445
Title: A Real-world Study: Efficacy and Safety of Eribulin in the Treatment of Advanced Breast Cancer
Brief Title: Efficacy and Safety of Eribulin in the Treatment of Advanced Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ying Wang, associate chief physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: 2020-KY-064
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; eribulin; real-world study
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; Trastuzumab; pertuzumab; pyrotinib; pembrolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HR+/HER2- advanced breast cancer: Efficacy and Safety of Eribulin in the Treatment of HR+/HER2- Advanced Breast Cancer
  Interventions: Drug: Eribulin
- HER2+ advanced breast cancer: Efficacy and Safety of Eribulin and anti-HER2 Targeted therapy in the Treatment of HER2+ advanced breast cancer
  Interventions: Drug: Eribulin; Drug: Trastuzumab; Drug: pertuzumab; Drug: Pyrotinib
- triple negative advanced breast cancer: Efficacy and Safety of Eribulin and Immunotherapy in the Treatment of triple negative advanced breast cancer
  Interventions: Drug: Eribulin; Drug: Pembrolizumab; Drug: Camerlizumab

INTERVENTIONS:
Drug: Eribulin — Eribulin，1.4mg/m2，Intravenous infusion，d1，d8，3-week cycle
  Other Names: Halaven
Drug: Trastuzumab — Trastuzumab，8mg/kg for the first dose，6mg/kg for the following dose，Intravenous infusion，3-week cycle
  Other Names: Herceptin
  Groups: HER2+ advanced breast cancer
Drug: pertuzumab — Pertuzumab，，840mg for the first dose，420mg for the following dose，Intravenous infusion，3-week cycle
  Other Names: Perjeta
  Groups: HER2+ advanced breast cancer
Drug: Pyrotinib — Pyrotinib，400mg，oral，every day
  Groups: HER2+ advanced breast cancer
Drug: Pembrolizumab — Pembrolizumab，200mg，Intravenous infusion，3-week cycle
  Other Names: Keytruda
  Groups: triple negative advanced breast cancer
Drug: Camerlizumab — Camerlizumab，200mg，Intravenous infusion，3-week cycle
  Groups: triple negative advanced breast cancer

SUMMARY:
Chemotherapy is an important means to prolong the survival time of advanced breast cancer. As a new type of microtubule inhibitor, eribulin has a unique mechanism of action. Compared with single drug chemotherapy, it can improve the overall survival time of 2.5 months, increase the clinical benefit rate by 5 times, and the tolerance of eribulin is good. Therefore, the guidelines at home and abroad recommend eribulin for the rescue of advanced breast cancer.

However, up to now, there is no large sample data on the efficacy of eribulin combined with anti HER2 targeted therapy in HER2 + metastatic breast cancer, and the efficacy of combined immunotherapy in triple negative metastatic breast cancer. Moreover, as a newly marketed chemotherapy drug in China, the efficacy and safety data of eribulin in Chinese population are relatively lacking. Therefore, we plan to include different types and line numbers of advanced breast cancer patients based on the Chinese population through real-world research, and receive the treatment regimen containing eribulin respectively. In HR + / her2-mbc, we use eribulin monotherapy; in HER2 + MBC, we use eribulin + anti HER2 targeted therapy; in TNBC, we use eribulin + immunotherapy / chemotherapy, The efficacy and safety of eribulin were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients (aged 18-80 years, including 18 and 80 years) with metastatic breast cancer confirmed by pathology or imaging are not suitable for surgical resection or radiotherapy for the purpose of cure;
2. The starting time of eribulin treatment was between January 2021 and December 2021;
3. They received no more than 2-line chemotherapy in the past;
4. In HR + / her2-mbc, patients were treated with eribulin monotherapy; in HER2 + MBC, patients were treated with eribulin + anti HER2 targeted therapy; in TNBC, patients were treated with eribulin + immunotherapy / chemotherapy; in patients with HER2 + MBC, patients were treated with eribulin + immunotherapy /chemotherapy;

Exclusion Criteria:

1. Patients without pathological diagnosis;
2. Patients with central nervous system metastasis;
3. She has received more than two chemotherapy regimens for metastatic breast cancer;
4. Participating in any intervention drug clinical trials.
5. Those who have been known to have allergic history to the components of this regimen;
6. The patient, the patient, or the person with serious harm to the safety of the study.
7. Any other situation in which the researcher considers that the patient is not suitable for the study may interfere with the concomitant diseases or conditions involved in the study, or there are any serious medical barriers that may affect the safety of the subjects (e.g., uncontrollable heart disease, hypertension, active or uncontrollable infection, active hepatitis B virus infection)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients (aged 18-80 years, including 18 and 80 years) with metastatic breast cancer confirmed by pathology or imaging are not suitable for surgical resection or radiotherapy for the purpose of cure
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival，PFS | up to 24 month
  The time from the beginning of treatment to the progression or death of the patient

SECONDARY OUTCOMES:
overall survival，OS | up to 36 month
  The time from the beginning of treatment to the death of the patient
Quality of life scale score，QoL | up to 24 month
  The quality of life score of patients during treatment was analyzed（FACT-B）. Performance Status Rating (PSR) was demonstrated for the FACT-B total score, which is the result of the following subscale scores: SWB (the Social / family Well-Being subscale) , EWB (the Emotional Well-Being subscale), AC (Additional Concerns subscale), PWB (the Physical Well-Being subscale), FWB (the Functional Well-Being subscale) Performance Status Rating (PSR) was demonstrated for the FACT-B total score, which is the result of the following subscale scores: SWB (the Social / family Well-Being subscale) , EWB (the Emotional Well-Being subscale), AC (Additional Concerns subscale), PWB (the Physical Well-Being subscale), FWB (the Functional Well-Being subscale)
Complete remission, CR | up to 12 month
  all target lesions disappeared, no new lesions appeared, and tumor markers were normal, which lasted for at least 4 weeks

OTHER OUTCOMES:
Partial remission, PR | up to 12 month
  the diameter of target lesions diminished more than 30% and lasted for 4 weeks
Disease stable, SD | up to 12 month
  the sum of the maximum diameter of the target lesion is smaller than PR, or the increase is not up to PD
Disease progression, PD | up to 12 month
  he sum of the maximum diameter of the target lesion increased by at least 20%, and its absolute value increased by at least 5 mm, New lesions are also considered as PD
Objective response rate , ORR | up to 12 month
  according to recist1.1 criteria, the proportion of patients whose best remission is CR or PR in the total number of evaluable patients.
Clinical benefit rate, CBR | up to 12 month
  according to recist1.1 criteria, the proportion of patients with Cr or PR or SD ≥ 24 weeks in the total number of evaluable patients.
Exploration of biomarkers | the first week after the enrollment
  Objective to explore the correlation between biomarkers and the ORR. The biomarkers will be test by nest-generation sequence, which include 520 genes and tumor mutation burden, like ERBB2/TP53/PIK3CA/ERBB4/CCND1 and so on.
the rate of adverse events | up to 24 month
  The probability and severity of adverse reactions were analyzed up to 2 year after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat Sen Memorial Hospital，Sun Yat sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacot W, Heudel PE, Fraisse J, Gourgou S, Guiu S, Dalenc F, Pistilli B, Campone M, Levy C, Debled M, Leheurteur M, Chaix M, Lefeuvre C, Goncalves A, Uwer L, Ferrero JM, Eymard JC, Petit T, Mouret-Reynier MA, Courtinard C, Cottu P, Robain M, Mailliez A. Real-life activity of eribulin mesylate among metastatic breast cancer patients in the multicenter national observational ESME program. Int J Cancer. 2019 Dec 15;145(12):3359-3369. doi: 10.1002/ijc.32402. Epub 2019 Jun 20. PMID 31087564
- [Result] Kimura K, Iwamoto M, Tanaka S, Yamamoto D, Yoshidome K, Ogura H, Terasawa R, Matsunami N, Takahashi Y, Nitta T, Morimoto T, Fujioka H, Kawaguchi K, Uchiyama K. A phase II, multicenter, single-arm trial of eribulin as first- or second-line chemotherapy for HER2-negative advanced or metastatic breast cancer: evaluation of efficacy, safety, and patient-reported outcomes. Cancer Chemother Pharmacol. 2018 May;81(5):923-933. doi: 10.1007/s00280-018-3567-y. Epub 2018 Mar 28. PMID 29594360
- [Result] Mayo-Wilson E, Heyward J, Keyes A, Reynolds J, White S, Atri N, Alexander GC, Omar A, Ford DE; National Clinical Trials Registration and Results Reporting Taskforce Survey Subcommittee. Clinical trial registration and reporting: a survey of academic organizations in the United States. BMC Med. 2018 May 2;16(1):60. doi: 10.1186/s12916-018-1042-6. PMID 29716585